CLINICAL TRIAL: NCT05392296
Title: Effects of Power Ball on Grip Strength in Children With Developmental Delay.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0703
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Developmental Delay
Keywords: power ball; Strengthening exercises; Hand grip; Developmental delay; Dynamometer
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Power ball (Experimental): experimental group getting the power ball training with conventional treatment
  Interventions: Other: Power ball; Other: isometric hand grip strengthening exercises
- Conventional (Active Comparator): group will be control group getting the conventional treatment (isometric hand grip training exercises)
  Interventions: Other: isometric hand grip strengthening exercises

INTERVENTIONS:
Other: Power ball — experimental group getting the power ball training with conventional treatment.
  Arms: Power ball
Other: isometric hand grip strengthening exercises — conventional treatment (isometric hand grip training exercises)

SUMMARY:
Developmental delay refers to the child who does not perform the normal milestones as other children accomplish in the same age within time or somehow late but can achieve them. While if the delay is found in two or more than two areas of the developmental skill it is known as Global Developmental Delay (GDD). It is divided into mild, moderate and severe developmental delay contributed by many other causes like prenatal, perinatal, postnatal and socioeconomic factors. The objective of the study is to determine the effects of power ball on grip strengthening children with developmental delay. In this study, we will randomly assigned 28 children into two groups, One group will be control group getting the conventional treatment (isometric hand grip training exercises) and other will be experimental group getting the power ball training with conventional treatment. During the sessions hand held dynamometer is use to check the grip strength. By using power ball grip strength in children with Developmental Delay can be improved.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-12 years
* Both genders (male /female)
* Moderate developmental delay
* Affected fine motor skill

Exclusion Criteria:

* With another neurological conditions(cerebral palsy, down's syndrome, Autism)
* Genetic disorder-

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Grip strength by Hand held Dynamometer | Baseline, 7th and 14th day
  A small portable device is held by the examiner and placed against the patient's limb during a maximal isometric contraction. A hand held dynamometer, however, takes the force a patient generates and transmits it through a transducer, quantifies the force, and then presents the data in a digital format. Health professionals can use this muscle strength testing equipment to measure muscle strength efficiently and effectively across the board. The purpose of using a hand dynamometer is to measure the maximum isometric strength of the hand and forearm muscles. The hand dynamometer can be adjusted for hand size and must be calibrated regularly for consistent results
Change in ABILHAND-KIDS tool scores | Baseline and 1 month
  The ABILHAND KIDS was originally developed by using the Rasch measurement model. It allows to convert ordinal score into linear measure located on unidimensional score.
  Procedure Parents are asked to fill the questionnaire according to child ability to do manual task ,ease in doing fine motor task and difficulty in performing activities, when the task are done1 Without other technical and human help(even if child actually uses help in daily life) 2 Irrespective of the limb actually used to do activity 3 Whatever strategy was used(any compensation is allowed

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Afzal, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Rising Sun Institute For Special Children, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choo YY, Agarwal P, How CH, Yeleswarapu SP. Developmental delay: identification and management at primary care level. Singapore Med J. 2019 Mar;60(3):119-123. doi: 10.11622/smedj.2019025. PMID 30997518
- [Background] Mithyantha R, Kneen R, McCann E, Gladstone M. Current evidence-based recommendations on investigating children with global developmental delay. Arch Dis Child. 2017 Nov;102(11):1071-1076. doi: 10.1136/archdischild-2016-311271. PMID 29054862
- [Background] Vitrikas K, Savard D, Bucaj M. Developmental Delay: When and How to Screen. Am Fam Physician. 2017 Jul 1;96(1):36-43. PMID 28671370
- [Background] Mussatto KA, Hoffmann RG, Hoffman GM, Tweddell JS, Bear L, Cao Y, Brosig C. Risk and prevalence of developmental delay in young children with congenital heart disease. Pediatrics. 2014 Mar;133(3):e570-7. doi: 10.1542/peds.2013-2309. Epub 2014 Feb 2. PMID 24488746
- [Background] Yoo S, Park SK, Yoon S, Lim HS, Ryu J. Comparison of Proprioceptive Training and Muscular Strength Training to Improve Balance Ability of Taekwondo Poomsae Athletes: A Randomized Controlled Trials. J Sports Sci Med. 2018 Aug 14;17(3):445-454. eCollection 2018 Sep. PMID 30116118